CLINICAL TRIAL: NCT06984744
Title: Effect of an Active Compound Containing Gum on Dental Plaque Formation on a 4-day Accumulation Model
Brief Title: 4-day Plaque Accumulation Model Evaluating Compound Containing Gum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lactea Therapeutics, LLC (Industry)
Collaborators: Indiana University (Other); Oral Health Research Institute, Indiana University School of Dentistry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LAC_IU_2025_plaque
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Dental Plaque Accumulation
Keywords: dental plaque; gum chewing
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Subjects who previously participated in other Oral Health Research Institute studies (OHRI) or who have contacted OHRI expressing interest in potential studies will be contacted by a team member who will conduct a screening phone interview. If the potential subjects appear to qualify, they will be scheduled for the screening visit.
  A sufficient number of subjects will be screened to participate, and 32 will be randomized to finish with at least 30 subjects. We intend to randomize a nearly equal number of female and male subjects. A unique screening number will identify all subjects screened for study participation. Screening numbers will be assigned according to appearance at the study site. Subjects who meet all inclusion and exclusion criteria will be randomized into the study. Block randomization will be used to assign subjects to one of the three treatment regimen sequences:
  1. Control regimen (Tx 3) followed by experimental regimen (Tx 1), followed by a negative control (Tx 2), or
Who Masked: Outcomes Assessor
Masking Description: The clinical examiners will remain blind to the individual subjects' treatment group during the study. If the treatment assignment must be unblinded for a subject, such as in the case of an emergency, the Principal Investigator will provide written documentation of the unblinding request. Otherwise, blinding will not be broken, unless required in the circumstances detailed above, until all subjects have completed the final study visit and the database has been monitored, locked, and approved by the Principal Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control regimen (No Intervention): Subjects will chew no gum during this regimen. Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Subjects in the no intervention regimen will use no gum. Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit.
- Intervention Experimental MIIP-E2 regimen (Experimental): Gum will contain gum base with 30mg of compound being evaluated. Gum will contain gum base only without compound being evaluated. Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit.
  Interventions: Device: MIIP-E2 containing gum
- Negative control regimen (Placebo Comparator): Gum will contain gum base only without compound being evaluated. Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit.
  Interventions: Device: placebo gum without MIIP-E2

INTERVENTIONS:
Device: MIIP-E2 containing gum — Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit. MIIP-E2 is an ultrapure (>99%) fully native and completely active form of bovine lactoferrin purified directly from raw milk.
  Arms: Intervention Experimental MIIP-E2 regimen
Device: placebo gum without MIIP-E2 — Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit.
  Arms: Negative control regimen

SUMMARY:
This will be a single-blind, single-center, 3-way crossover, randomized controlled clinical trial with 3 treatment periods utilizing 32 subjects. (Fig 1, in protocol) Each treatment period will be 4 days (96 hours +/-3 hours) in accordance with the plaque accumulation model using one of the following treatment groups: an active compound MIIP-E2 gum (experimental regimen), an inactive compound gum (negative control regimen), and a no-gum (control regimen).

DETAILED DESCRIPTION:
treatment periods utilizing 32 subjects. (Fig 1, in protocol) Each treatment period will be 4 days (96 hours +/-3 hours) in accordance with the plaque accumulation model using one of the following treatment groups: an active compound MIIP-E2 gum (experimental regimen), an inactive compound gum (negative control regimen), and a no-gum (control regimen). Each subject will be assigned to one of the following three treatment regimen sequences:

1. Control regimen followed by experimental regimen, followed by a negative control regimen, or
2. Experimental regimen followed by negative control regimen, followed by control regimen or
3. Negative control regimen followed by control regimen, followed by an experimental regimen Subjects will be asked to refrain from oral hygiene (OH) procedures and chewing gum 12 hours (+/- 2 hours) and from eating or drinking (except for water) 2 hours prior to the screening visit. During the 4-day study treatment periods, subjects will also be asked to refrain from oral hygiene practices or any elective dental treatment. Subjects can resume their regular oral hygiene procedures during the wash-out periods of approximately 10 days.

At the screening, potential subjects will be given the IRB (Institutional Review Board)-approved informed consent form to read and ask questions. Also, adequate time to decide about their participation will be provided. A study representative trained and delegated by the Principal Investigator will review the IRB-approved consent and answer any questions the potential subject might have before the subject signs/dates the consent. After the subject signs and dates the consent, the study representative will sign and date the consent to confirm that the consent process was completed before initiating any study procedures. The subject will be given a copy of the signed/dated consent.

A designated staff member will collect the medical and concomitant medication information for the study dentist's review. The dentist will perform an oral examination and a PLI to assess the subject's whole-mouth plaque accumulation. A score of 2 or greater will be needed to comply with the study inclusion criteria based on the Turesky modification of the Quigley and Hein Plaque Index (PLI). Other dental characteristics specified on the inclusion/ exclusion criteria will be assessed to determine study eligibility. Eligible subjects will receive a dental prophylaxis and be scheduled for a baseline appointment.

During the baseline appointment, the subjects' continuance criteria and OST (oral specimen test) examination will be assessed, and an unstimulated saliva sample will be collected. Subjects' teeth will be polished, flossed, and subsequently stained to evaluate total plaque removal and an oral assessment will be performed to confirm the complete removal of plaque. If any plaque is found, the plaque will be removed by either flossing, repolishing the surface, or with an instrument. The dental examiner will assess PLI. Intraoral photos will be taken, including one front and two lateral images (right and left side). 32 subjects will be enrolled and randomly assigned to one of the treatment regimens. Subjects assigned to experimental and negative treatment regimens will perform the first product use under supervision.

Each subject will be instructed to refrain from using any oral dental hygiene procedures during the study treatment period (4 days). Subjects assigned to the experimental and negative treatment regimen will use only the provided gum product three times a day for 10 minutes after meals (breakfast, lunch, and dinner). Starting on one side of the mouth, chewing for 1 minute, and switching to the other side for another minute. Afterward, they continue chewing for the remaining time however they like. To assess compliance, each subject assigned to a chewing gum product will be provided a diary to record every time they use the product and record any events associated with their study participation. Finally, subjects will be scheduled to return for an end-of-regimen visit.

The last product-use treatment will be after dinner the day before the visit. Subjects will refrain from eating or drinking (except water) for two hours before their appointment. They will also be asked to rinse their mouths with water approximately 30 minutes before their visit.

During the end of the treatment visit, subjects' continuance criteria will be assessed; the diary will be reviewed for compliance; an OST exam will be performed; and an unstimulated saliva sample will be collected. Subjects will rinse with a disclosing solution to reveal the accumulation of dental plaque. Intraoral photos, including one front and two lateral images (right and left sides), will be taken. Afterward, the examiner will assess the PLI, and subjects will be taken to a brushing station to brush their teeth using a provided toothbrush, fluoride-containing toothpaste, and dental floss. They will be scheduled for the next visit after a washout period of approximately 10 days.

For treatments 2 and 3, the procedures mentioned in the baseline visit will be repeated (except for randomization). A new product (or no product) will be given according to the randomization assignment. The end of the treatment visit will be repeated on the fourth day of each treatment period.

Lactea Therapeutics has formulated a gum product containing an active innate immune protein, MIIP-E2. This product is an ultrapure (>99%) fully native and completely active form of bovine lactoferrin extracted and purified directly from raw milk. MIIP-E2 aims to develop a field-deployable dental care solution to enhance on-the-go oral care targeting military use. Due to the capability of the MIIP-E2 gum to coat the inner surfaces of the mouth, it can function as a barrier to biofilm adherence. The dosage of MIIP-E2 proposed for use in this study is dramatically below these acceptable levels in milk-based infant formulas, which range between 101.3 and 60.1 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between 18 and 65 years old
* Willing to read and sign the IRB-approved informed consent.
* Healthy, as determined by pertinent medical history at the study dentist's discretion.
* A minimum of 20 natural teeth (excluding third molars) with at least two scorable surfaces per tooth (teeth with full crowns, large/extensive restorations on the interproximal areas, and orthodontic bands will not be included in the tooth count)
* PLI of 2 or greater (Based on the Turesky modification of the Quigley and Hein Plaque Index) calculation based on a whole mouth plaque score.
* Willing to comply with the study procedures.

Exclusion Criteria:

* Presence of any acute or chronic condition, organ system disease, or medication that, in the principal investigator's opinion, could compromise the subjects' ability to participate in the study.
* Gross oral pathologies, including caries, calculus, or soft tissue conditions that show evidence of chronic neglect.
* Evidence of acute periodontal conditions or periodontitis with pockets greater than 5 mm on more than one site
* Use of antibiotics 30 days prior to or during the study
* Requiring the need for antibiotic premedication prior to dental procedures
* Sensitivity to bovine products (lactoferrin) or any of the listed inactive ingredients
* Orthodontic appliances or any removable, except lingual bar retainers
* Self-reported pregnant, wanting to get pregnant, or breast-feeding female,
* Self-reported allergy to disclosing solution ingredients (red dye #28)
* Acute Temporomandibular Disorders (TMD)
* Subject who has participated in other studies (including non-medicinal studies) involving product(s) within 30 days before study screening.
* Subject who has previously been randomized in this study
* An employee of the study site directly involved with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
dental plaque | At the end of 4 days of intervention.
  Dental plaque was identified using a disclosing solution and scored using the Turesky modification of the Quigley-Hein Plaque Index (PLI). The index score was scored between 0 and 5, with 0 = no plaque detected and 5= = Plaque covering 2/3 or more of the tooth's crown. The remaining values are based on the amount of plaque covering the tooth. The higher the score, the more plaque accumulated and the worse the outcome for the surface. Each tooth, except the third molars, will be scored at six sites: Mesio-Buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual. The plaque score index for an individual is determined by adding all the individual scores and dividing the total score by the number of surfaces examined. A score would range from 0.1 to 3.0 (0.1-1.0= = mild inflammation; 1.1-2.0= = moderate inflammation; and 2.1-3.0= = severe inflammation).

SECONDARY OUTCOMES:
16S sequencing | At the end of 4 days of intervention.
  In addition, patient saliva samples will be taken before and after each treatment regimen for 16S rRNA (ribosomal ribonucleic acid) microbiome sequencing using the Qiagen PAXgene Saliva Collector and protocols that accompany the collection kit (https://www.qiagen.com /us/products/discovery-and-translational-research/sample-collection-stabilization/dna/pax gene-saliva-collector). Sequencing will be performed at CD Genomics (a third-party vendor) using protocols for full-length PacBio (Pacific Biosciences) sequencing and IRB#: 25945 Version Date: February 3, 2025 Page 6 of 18 analyzed using standard methodologies to identify microbial taxonomy. No human genetic information will be collected or analyzed using this methodology.
Dental Plaque Visual Assessment with photographs | At the end of 4 days of intervention.
  Images of dental plaque will be used for both qualitative representations of outcomes in future reports as well as used as a secondary, complementary quantitative analysis for the PLI assessment. For the quantitative analysis, plaque coverage on teeth will be assessed using an image thresholding area measurement as previously described. This analysis is anticipated to provide similar results to the PLI as mentioned earlier but may allow for further analysis and quantitative precision. Depending on preliminary analysis, these measurements may be used to further assess details of product efficacy, such as regional changes in plaque across teeth, to understand whether the reduction in plaque occurred primarily on surfaces with direct exposure to the gum or throughout the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Ana G Gossweiler, DDMSD, Principal Investigator — Oral Health Research Institute Indiana University
Locations (1):
- Oral Health Research Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Claydon NC, Hall C, Hughes AJ, Shaw D, Seong J, Davies M, West NX. Randomized controlled trial to study plaque inhibition in calcium sodium phosphosilicate dentifrices. J Dent. 2016 Mar;46:61-7. doi: 10.1016/j.jdent.2016.01.003. Epub 2016 Jan 12. PMID 26796897
- [Result] Smith RN, Brook AH, Elcock C. The quantification of dental plaque using an image analysis system: reliability and validation. J Clin Periodontol. 2001 Dec;28(12):1158-62. doi: 10.1034/j.1600-051x.2001.281211.x. PMID 11737514
- [Result] Buetas E, Jordan-Lopez M, Lopez-Roldan A, D'Auria G, Martinez-Priego L, De Marco G, Carda-Dieguez M, Mira A. Full-length 16S rRNA gene sequencing by PacBio improves taxonomic resolution in human microbiome samples. BMC Genomics. 2024 Mar 25;25(1):310. doi: 10.1186/s12864-024-10213-5. PMID 38528457
- [Result] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Result] Morita Y, Ishikawa K, Nakano M, Wakabayashi H, Yamauchi K, Abe F, Ooka T, Hironaka S. Effects of lactoferrin and lactoperoxidase-containing food on the oral hygiene status of older individuals: A randomized, double blinded, placebo-controlled clinical trial. Geriatr Gerontol Int. 2017 May;17(5):714-721. doi: 10.1111/ggi.12776. Epub 2016 May 6. PMID 27150460
- [Result] Nakano M, Yoshida A, Wakabayashi H, Tanaka M, Yamauchi K, Abe F, Masuda Y. Effect of tablets containing lactoferrin and lactoperoxidase on gingival health in adults: A randomized, double-blind, placebo-controlled clinical trial. J Periodontal Res. 2019 Dec;54(6):702-708. doi: 10.1111/jre.12679. Epub 2019 Jul 10. PMID 31292969
- [Result] Arslan SY, Leung KP, Wu CD. The effect of lactoferrin on oral bacterial attachment. Oral Microbiol Immunol. 2009 Oct;24(5):411-6. doi: 10.1111/j.1399-302X.2009.00537.x. PMID 19702956
- [Result] Velusamy SK, Markowitz K, Fine DH, Velliyagounder K. Human lactoferrin protects against Streptococcus mutans-induced caries in mice. Oral Dis. 2016 Mar;22(2):148-54. doi: 10.1111/odi.12401. Epub 2016 Jan 18. PMID 26601919
- [Result] Berlutti F, Pilloni A, Pietropaoli M, Polimeni A, Valenti P. Lactoferrin and oral diseases: current status and perspective in periodontitis. Ann Stomatol (Roma). 2011 Mar;2(3-4):10-8. Epub 2012 Jan 27. PMID 22545184
- [Result] Yamauchi K, Toida T, Nishimura S, Nagano E, Kusuoka O, Teraguchi S, Hayasawa H, Shimamura S, Tomita M. 13-Week oral repeated administration toxicity study of bovine lactoferrin in rats. Food Chem Toxicol. 2000 Jun;38(6):503-12. doi: 10.1016/s0278-6915(00)00036-3. PMID 10828502
- [Result] Cao X, Ren Y, Lu Q, Wang K, Wu Y, Wang Y, Zhang Y, Cui XS, Yang Z, Chen Z. Lactoferrin: A glycoprotein that plays an active role in human health. Front Nutr. 2023 Jan 5;9:1018336. doi: 10.3389/fnut.2022.1018336. eCollection 2022. PMID 36712548
- [Result] Drago-Serrano ME, de la Garza-Amaya M, Luna JS, Campos-Rodriguez R. Lactoferrin-lipopolysaccharide (LPS) binding as key to antibacterial and antiendotoxic effects. Int Immunopharmacol. 2012 Jan;12(1):1-9. doi: 10.1016/j.intimp.2011.11.002. Epub 2011 Nov 18. PMID 22101278
- [Result] Smith AJ, Moran J, Dangler LV, Leight RS, Addy M. The efficacy of an anti-gingivitis chewing gum. J Clin Periodontol. 1996 Jan;23(1):19-23. doi: 10.1111/j.1600-051x.1996.tb00499.x. PMID 8636452
- [Result] Weber J, Scholz KJ, Schenke IM, Pfab F, Cieplik F, Hiller KA, Buchalla W, Sahm C, Kirschneck C, Paddenberg-Schubert E. Randomized controlled clinical trial on the efficacy of a novel antimicrobial chewing gum in reducing plaque and gingivitis in adolescent orthodontic patients. Clin Oral Investig. 2024 Apr 25;28(5):272. doi: 10.1007/s00784-024-05669-4. PMID 38664261
- [Result] Takenouchi A, Saeki Y, Otani E, Kim M, Fushimi A, Satoh Y, Kakegawa Y, Arai H, Taguchi N, Matsukubo T. Effects of Chewing Gum Base on Oral Hygiene and Mental Health: A Pilot Study. Bull Tokyo Dent Coll. 2021 Mar 13;62(1):7-14. doi: 10.2209/tdcpublication.2020-0009. Epub 2021 Feb 15. PMID 33583877
- [Result] Dodds MW. The oral health benefits of chewing gum. J Ir Dent Assoc. 2012 Oct-Nov;58(5):253-61. PMID 23573702
- [Result] Crystal YO, Luo YL, Duangthip D, Tantawi ME, Benzian H, Schroth RJ, Feldens CA, Virtanen JI, Al-Batayneh OB, Diaz ACM, Vukovic A, Pavlic V, Mfolo T, Daryanavard HA, Gaffar BO, Shamala A, Folayan MO; Early Childhood Caries Advocacy Group (ECCAG). A scoping review of the links between early childhood caries and clean water and sanitation: the Sustainable Development Goal 6. BMC Oral Health. 2024 Jul 9;24(1):769. doi: 10.1186/s12903-024-04535-9. PMID 38982426
- [Result] Devinsky O, Boyce D, Robbins M, Pressler M. Dental health in persons with disability. Epilepsy Behav. 2020 Sep;110:107174. doi: 10.1016/j.yebeh.2020.107174. Epub 2020 Jun 9. PMID 32531727
- [Result] Chiappelli F, Bauer J, Spackman S, Prolo P, Edgerton M, Armenian C, Dickmeyer J, Harper S. Dental needs of the elderly in the 21st century. Gen Dent. 2002 Jul-Aug;50(4):358-63. PMID 12640853
- [Result] Milleman K, Milleman J, Bosma ML, McGuire JA, Sunkara A, DelSasso A, York T, Cecil AM. Role of Manual Dexterity on Mechanical and Chemotherapeutic Oral Hygiene Regimens. J Dent Hyg. 2022 Jun;96(3):35-45. PMID 35654566
- [Result] Salzer S, Graetz C, Dorfer CE, Slot DE, Van der Weijden FA. Contemporary practices for mechanical oral hygiene to prevent periodontal disease. Periodontol 2000. 2020 Oct;84(1):35-44. doi: 10.1111/prd.12332. PMID 32844413
- [Result] Ruiz Nunez MDR, da Luz Raulino M, Goulart Castro R, Schaefer Ferreira de Mello AL. Dental plaque control strategies for the elderly population: A scoping review. Int J Dent Hyg. 2022 Feb;20(1):167-181. doi: 10.1111/idh.12497. Epub 2021 Apr 14. PMID 33829631
- [Result] Sanz M, Beighton D, Curtis MA, Cury JA, Dige I, Dommisch H, Ellwood R, Giacaman RA, Herrera D, Herzberg MC, Kononen E, Marsh PD, Meyle J, Mira A, Molina A, Mombelli A, Quirynen M, Reynolds EC, Shapira L, Zaura E. Role of microbial biofilms in the maintenance of oral health and in the development of dental caries and periodontal diseases. Consensus report of group 1 of the Joint EFP/ORCA workshop on the boundaries between caries and periodontal disease. J Clin Periodontol. 2017 Mar;44 Suppl 18:S5-S11. doi: 10.1111/jcpe.12682. PMID 28266109
- [Result] Arweiler NB, Netuschil L. The Oral Microbiota. Adv Exp Med Biol. 2016;902:45-60. doi: 10.1007/978-3-319-31248-4_4. PMID 27161350

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT06984744/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT06984744/ICF_001.pdf